CLINICAL TRIAL: NCT01278264
Title: Transversus Abdominis Plane Blocks in Patients Scheduled for an Abdominoplasty. A Prospective, Randomized, Double Blind, Comparison Between the Posterior Approach and Placebo.
Brief Title: Transversus Abdominis Plane Blocks With Abdominoplasty
Acronym: TAPA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinique Saint-Jean, Bruxelles (Other)
Responsible Party: Arnaud G Bosteels, Service Anesthesie Clinique Saint-Jean Bruxelles
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: ANESAB001
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-02

CONDITIONS: Post Operative Pain
Keywords: Transversus abdominis plane block; Ultrasound guided; Abdominoplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- iTAP-group (Active Comparator): Posterior approach for TAP: ultrasound guided bilateral needle insertion in the transversus abdominis plane, anterior to the quadratus lumborum muscle
  Interventions: Drug: Ropivacaine 0.25%, 0.5 ml/kg
- aTAP-group (Active Comparator): Subcostal approach for TAP: US guided needle insertion in the transversus abdominis plane, lateral to rectus sheet
  Interventions: Drug: Ropivacaine 0.25%, 0.5 ml/kg

INTERVENTIONS:
Drug: Ropivacaine 0.25%, 0.5 ml/kg — Posterior approach for TAP: ultrasound guided bilateral needle insertion in the transversus abdominis plane, anterior to the quadratus lumborum muscle
  Arms: iTAP-group
Drug: Ropivacaine 0.25%, 0.5 ml/kg — Subcostal approach for TAP: US guided needle insertion in the transversus abdominis plane, lateral to rectus sheet
  Arms: aTAP-group

SUMMARY:
Comparing morphine consumption and recovery with two different TAP block techniques after abdominoplasty.

DETAILED DESCRIPTION:
TAP blocks have the potential to become an important part of multi-modal analgesia after abdominal surgery (1,2). Originally Dr J McDonnell described a blind double pop technique, trough the triangle of Petit, with up to 48 hours of analgesia (3,4). Dr P Hebbard described an ultrasound based technique with a subcostal (for supra-umbilical analgesia) and an axillary mid-line injection (for sub-umbilical analgesia) in the TAP, with reported analgesia for up to 8 hours (5,6). Recently Dr J McDonnell presented data showing para vertebral spread (up to L5) of the (high dose, low concentration) local anaesthetic explaining the prolonged analgesic effect (7,8). In 2007 Dr Blanco described an ultrasound guided technique for the posterior inﬁltration as performed by McDonnell (9). Our limited observational comparison between both block techniques conﬁrms this difference. We decided to compare both techniques (the ultrasound guided single shot subcostal injection, the aTAP-group (Hebbard is from Australia) and the ultrasound guided posterior injection, the iTAP-group (McDonnell is from Ireland). We will use the same volume and concentration of local anesthetic and we will asses their analgesic efﬁcacy and improvement in quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for abdominoplasty
* ASA 1-2
* Fluent french/dutch/english

Exclusion Criteria:

* History of allergy to local anaesthetics
* Chronic opioids abuse
* Pregnant patients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-05 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | 48 hours
  Consumption measured by the use of the PCA pump

SECONDARY OUTCOMES:
VAS score | 48 hours
Post operative nausea and vomiting | 48 hours
Constipation | 48 hours
Pruritus | 48 hours
First time to get up | 48 hours
First time to eat | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud G Bosteels, MD, Principal Investigator — Clinique Saint-Jean, Bruxelles
Locations (1):
- Clinique Saint Jean, Brussels, Belgium

REFERENCES:
- [Background] Charlton S, Cyna AM, Middleton P, Griffiths JD. Perioperative transversus abdominis plane (TAP) blocks for analgesia after abdominal surgery. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD007705. doi: 10.1002/14651858.CD007705.pub2. PMID 21154380
- [Background] Petersen PL, Mathiesen O, Torup H, Dahl JB. The transversus abdominis plane block: a valuable option for postoperative analgesia? A topical review. Acta Anaesthesiol Scand. 2010 May;54(5):529-35. doi: 10.1111/j.1399-6576.2010.02215.x. Epub 2010 Feb 17. PMID 20175754
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] 6. McDonnell J. XXIX Annual ESRA congress - Porto, Portugal, 2010.
- [Background] 7. Blanco R. TAP block under ultrasound guidance: the description of a
- [Background] Griffiths JD, Barron FA, Grant S, Bjorksten AR, Hebbard P, Royse CF. Plasma ropivacaine concentrations after ultrasound-guided transversus abdominis plane block. Br J Anaesth. 2010 Dec;105(6):853-6. doi: 10.1093/bja/aeq255. Epub 2010 Sep 22. PMID 20861094
- [Background] Ingrande J, Lemmens HJ. Dose adjustment of anaesthetics in the morbidly obese. Br J Anaesth. 2010 Dec;105 Suppl 1:i16-23. doi: 10.1093/bja/aeq312. PMID 21148651
- [Background] 5. McDonnell J. Ultrasound guided abdominal wall blocks. X Annual BARA meeting -Brussels, Belgium, 2010
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039